CLINICAL TRIAL: NCT05454943
Title: Proof-of-Concept of Time-Restricted Eating as a Novel Lifestyle Intervention for Breast Cancer Prevention
Brief Title: Remote Time-restricted EAting DeliverY
Acronym: READY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Amy Kirkham, Amy Kirkham, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIS42756
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Disturbance
MeSH Terms: interventions — Trehalase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Standardized TRE protocol + External Support (Experimental): Participants will be asked to follow a standardized 16:8 TRE protocol with an 11 am to 7 pm eating window for 16 weeks. Participants receive support to follow the TRE intervention from the study team which will include an initial consultation with a registered dietitian and ongoing tailored feedback via brief support calls from study staff at weeks 1, 3, 6, and 12.
  Interventions: Behavioral: Standardized TRE Protocol; Behavioral: External Support for TRE
- Standardized TRE protocol + Peer Support (Experimental): Participants will be asked to follow a standardized 16:8 TRE protocol with an 11 am to 7 pm eating window for 16 weeks. Each participant will be matched with another participant in the same group to provide peer-based support to adhere to TRE. Study staff will introduce pairs and provide an introduction to TRE and then pairs will meet by phone/video at weeks 1, 3, 6, and 12 at a minimum, with additional contact encouraged.
  Interventions: Behavioral: Standardized TRE Protocol; Behavioral: Peer Support for TRE
- Personalized TRE protocol + External Support (Experimental): Participants will be asked to follow TRE for 16 weeks with a protocol that is personalized to their preferences within the following pre-specified rules: 1) 8-10 hour eating window; 2) self-selected eating window start time as long as it ends ≥3h before bedtime; 3) if days off are required, aim to do so after following TRE for ≥5 successive days each week. Participants receive support to follow the TRE intervention from the study team which will include an initial consultation with a registered dietitian and ongoing tailored feedback via brief support calls from study staff at weeks 1, 3, 6, and 12.
  Interventions: Behavioral: Personalized TRE Protocol; Behavioral: External Support for TRE
- Personalized TRE protocol + Peer Support (Experimental): Participants will be asked to follow TRE for 16 weeks with a protocol that is personalized to their preferences within the following pre-specified rules: 1) 8-10 hour eating window; 2) self-selected eating window start time as long as it ends ≥3h before bedtime; 3) if days off are required, aim to do so after following TRE for ≥5 successive days each week. Each participant will be matched with another participant in the same group to provide peer-based support to adhere to TRE. Study staff will introduce pairs and provide an introduction to TRE and then pairs will meet by phone/video at weeks 1, 3, 6, and 12 at a minimum, with additional contact encouraged.
  Interventions: Behavioral: Personalized TRE Protocol; Behavioral: Peer Support for TRE
- Control Group (No Intervention): Participants will be asked to maintain their usual diet and physical activity patterns for 16 weeks. They will receive the same number and timing of calls from study staff as the other groups (at randomization, 1, 3, 6, 12 weeks).

INTERVENTIONS:
Behavioral: Standardized TRE Protocol — A standardized 16:8 TRE protocol with an 11 am to 7 pm eating window.
  Arms: Standardized TRE protocol + External Support; Standardized TRE protocol + Peer Support
Behavioral: Personalized TRE Protocol — A personalized TRE protocol following pre-specified rules: 1) 8-10 hour eating window; 2) self-selected eating window start time as long as it ends ≥3h before bedtime; 3) if days off are required, aim to do so after following TRE for ≥5 successive days each week.
  Arms: Personalized TRE protocol + External Support; Personalized TRE protocol + Peer Support
Behavioral: External Support for TRE — External support (from study staff) that includes consultation with a registered dietitian and ongoing tailored feedback via support calls at weeks 1, 3, 6, and 12.
  Arms: Personalized TRE protocol + External Support; Standardized TRE protocol + External Support
Behavioral: Peer Support for TRE — Matched pairs will meet by phone/video at weeks 1, 3, 6, and 12.
  Arms: Personalized TRE protocol + Peer Support; Standardized TRE protocol + Peer Support

SUMMARY:
This study will evaluate the implementation and effectiveness of free-living TRE on biological and behavioural breast cancer risk factors.

DETAILED DESCRIPTION:
TRE is an eating pattern where individuals consume ad libitum energy intake within a set window of time, commonly 8 hours, which induces a fasting window of 16 hours per day (i.e., 16:8 TRE). TRE is a simple and accessible lifestyle intervention with high adherence potential that may target both biological and behavioural mechanisms of breast cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* Females
* No cancer history
* ≥50 years old
* Have metabolic dysfunction (defined as self-reported diagnosis of pre-diabetes, type 2 diabetes, or at least moderate Canadian diabetes risk (CANRISK) score)
* Access to an Ontario Lifelabs location
* Owns a smartphone with Bluetooth capability with Apple or Android operating system

Exclusion Criteria:

* Type 1 diabetes
* Taking exogenous insulin, sulfonylureas, or GLP-1 receptor agonists
* Self-reported history of an eating disorder
* BMI <18.5 kg/m
* Working night or rotating shifts
* Eating window <12 hours or consistently eating less than 3 meals/day in the past 3 months
* Major dietary changes within the past 3 months (i.e. calorie counting, ketogenic diet)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Adherence to TRE for the 16-week intervention | 16-week average
  Assessed daily through twice daily automated text messages asking participants to respond with what time they started and stopped eating that day.
Hemoglobin A1c | 16 Weeks
  Collected via venipuncture

SECONDARY OUTCOMES:
HOMA-IR | 16 Weeks
  Homeostatic Model Assessment for Insulin Resistance calculated as fasting glucose in mmol/l*fasting insulin in μU/ml/22.5
Free-living glucose control | 16 Weeks
  Participants will be provided with a Dexcom G6 continuous glucose monitor transmitter and sensor. This data will be evaluated as the 5-day average of: 24-hour, daytime, and nocturnal glucose concentration, time in hyper, normo and hypoglycemia, and glycemic variability
C-Reactive Protein | 16 Weeks
  Measured via venipuncture and core lab lab analysis
Lipid profile | 16 Weeks
  Measured via venipuncture and core lab lab analysis
Body weight | 16 Weeks
  Measured via Fitbit Aria Air scale at baseline and 16-weeks but also once per week to evaluate trajectory of change
Waist circumference | 16 weeks
  Measured via provided circumference measuring tape as the average of 2 measurements
Blood Pressure | 16 Weeks
  Participant will be provided with a Bios 3al1-3e blood pressure measuring device. After 5 minutes of quiet seated rest, blood pressure will be measured 6 times, 60 seconds apart in a standardized seated position with the average of the 2nd through 6th measurement used.
10-year cardiovascular disease risk | 16 Weeks
  Calculated via both the Framingham and Reynolds 10-year CVD risk scores using measured collected for study purposes (i.e., age, total cholesterol, HDL, systolic blood pressure, smoking status, C-reactive protein, family history of heart disease).
Metabolic syndrome (NCEP/ATP III criteria) | 16 Weeks
  As defined by the NCEP/ATP III criteria using measurements taken using provided study tools
Metabolic syndrome z-score | 16 Weeks
  As defined by the NCEP/ATP III criteria and age and ethnic specific calculations
Alanine Aminotransferase | 16 Weeks
  Measured via venipuncture and core lab lab analysis
TRE acceptability and appropriateness | 16 Weeks
  Evaluated via an 'End of Study Survey' (including a Diet Satisfaction Score Tool and acceptability questions) and semi-structured qualitative interviews
TRE Adoption | 16 Weeks
  Evaluated as uptake of each delivery model, defined as adherence to the intervention touch points (i.e., external support: support calls with staff; peer support: number of peer interactions; both: response rate to adherence).
Cost of intervention delivery | 16 Weeks
  Intervention costs will be evaluated and averaged per participant from the time required for intervention phone calls, scheduling, and technical support for adherence app by the study staff according to hourly rates of pay.
TRE Sustainability | 1, 2, 3, and 4 months post intervention period
  Evaluated via participant self-report of continued TRE post-intervention
TRE Adverse Events | 16 Weeks
  Measured via experience of selected relevant Common Terminology Criteria for Adverse Events (CTCAE v5) with additional questions about duration and change in the revised 18-item version of the Three-Factor Eating Questionnaire (aka Eating Inventory)
Health-related quality of life | 16 Weeks
  Measured by the RAND-36 Physical Component Summary. Physical component summary of the RAND-36 questionnaire (minimum = 0, maximum = 50, a higher score is a better outcome)
Sleep duration | 16 Weeks
  Measured via FitBit Inspire 2 as 7-day average
Sedentary time | 16 Weeks
  Measured via FitBit Inspire 2 as 7-day average
Physical activity | 16 Weeks
  Measured via FitBit Inspire 2 as 7-day average

OTHER OUTCOMES:
Anxiety | 16 weeks
  Evaluated via the Hospital Anxiety and Depression Scale (HADS); This 14-item questionnaire has a minimum score of 0 and maximum of 21, where a higher score is worse.
Depression | 16 weeks
  Evaluated via the Hospital Anxiety and Depression Scale (HADS); This 14-item questionnaire has a minimum score of 0 and maximum of 21, where a higher score is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Kirkham, PhD, Principal Investigator — University of Toronto
Locations (1):
- Remote Ontario-wide, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No